CLINICAL TRIAL: NCT05473598
Title: Stand Down-Think Before You Drink: An RCT of a Mobile App for Hazardous Drinking With Peer Phone Support
Acronym: PS-Stand Down
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 20-093
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Alcoholism
Keywords: Alcohol use disorder; Mobile health; Peer Support
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual Care (Active Comparator): All patients, regardless of condition, will have access to usual care for hazardous drinking in primary care. In this setting, usual care entails a spectrum of alcohol-related services including annual screening for hazardous drinking, brief intervention following a positive screen (advice from a provider to reduce their drinking), and referral (as needed) to specialty AUD treatment.
  Interventions: Behavioral: Stand Down app; Behavioral: Peer-Supported Stand Down; Other: Usual Care
- UC + Stand Down app (app only) (Experimental): Patients in this condition will receive Usual Care (UC) and be provided a unique code and password to access Stand Down. The app is based on principles of motivational enhancement and cognitive-behavioral therapies and comprises 7 modules organized around 4 goals: 7 modules organized around 4 goals: (i) Enhance awareness of drinking patterns (assessment and personalized feedback), (ii) Establish and monitor progress towards drinking goal - i.e., moderation or abstinence, (iii) Manage cravings and other problems using in-the-moment tools, and (iv) Connect users with other types of support. App usage will be tracked by the research team for the duration of the study (32 weeks).
  Interventions: Behavioral: Stand Down app; Behavioral: Peer-Supported Stand Down
- UC + Peer-Supported Stand Down (PS-Stand Down) (Experimental): Patients assigned to this condition will receive UC and access to Stand Down, plus four phone sessions from a Peer over 8 weeks. Sessions will be bi-weekly, approximately 15-30 minutes in length, and focus on enhancing patients' engagement with the app.
  Interventions: Behavioral: Peer-Supported Stand Down

INTERVENTIONS:
Behavioral: Stand Down app — Patients in this condition will receive Usual Care (UC) and be provided a unique code and password to access Stand Down. The app is based on principles of motivational enhancement and cognitive-behavioral therapies and comprises 7 modules organized around 4 goals: 7 modules organized around 4 goals: (i) Enhance awareness of drinking patterns (assessment and personalized feedback), (ii) Establish and monitor progress towards drinking goal - i.e., moderation or abstinence, (iii) Manage cravings and other problems using in-the-moment tools, and (iv) Connect users with other types of support. App usage will be tracked by the research team for the duration of the study (32 weeks).
  Other Names: App only
  Arms: UC + Stand Down app (app only); Usual Care
Behavioral: Peer-Supported Stand Down — Patients assigned to this condition will receive UC and access to Stand Down, plus four phone sessions from a Peer over 8 weeks. Sessions will be bi-weekly, approx. 15-30 minutes in length, and focus on enhancing patients' engagement with the app.
  Other Names: PS-Stand Down
Other: Usual Care — All patients, regardless of condition, will have access to usual care for hazardous drinking in primary care. In this setting, usual care entails a spectrum of alcohol-related services including annual screening for hazardous drinking, brief intervention following a positive screen (advice from a provider to reduce their drinking), and referral (as needed) to specialty AUD treatment.
  Other Names: UC
  Arms: Usual Care

SUMMARY:
Hazardous drinking is common among Veteran primary care patients and increases risk for more costly and complex medical problems over the long-term. Yet, the vast majority of these Veterans go untreated. By providing an option for care that is easily accessible, private, and self-directed, mobile applications (apps) circumvent many barriers to alcohol use treatment. However, poor patient engagement remains the Achilles' heel of these apps. Through supportive accountability, Peer Specialists can maximize the reach and engagement of these apps with patients and improve drinking outcomes. The goal of this project is to evaluate whether an app for alcohol use self-management ("Stand Down") reduces drinking among Veteran primary care patients who engage in hazardous drinking, and for whom Peer-Supported-Stand Down is more effective than the app alone. If successful, the proposed research has the potential to transform care and increase access to alcohol-related services for Veterans who engage in hazardous drinking but rarely seek treatment, and, in turn, mitigate the adverse health outcomes that stem from untreated hazardous drinking.

DETAILED DESCRIPTION:
One in four Veterans presenting to VA primary care screen positive for hazardous drinking. However, due to barriers such as Veterans' stigma about seeking alcohol use treatment and challenges with traveling to VA, most of these Veterans do not receive any alcohol-related care. Mobile applications (apps) are an innovative means of expanding access to alcohol use treatment. The evidence for mobile apps, such as "Step Away", to improve drinking outcomes is emerging. Nevertheless, poor patient engagement remains the Achilles' heel of these apps. Peer Specialists ("Peers") can facilitate Veterans' engagement with mobile apps intended for self-management of hazardous drinking by helping to orient patients to these apps and by providing technical support and accountability. In a VA HSR&D pilot study, the investigators created a Veteran version of the Step Away app ("Stand Down: Think Before You Drink") and conducted an open trial in which Veterans with hazardous drinking used the app while receiving Peer phone support. The intervention ("Peer-Supported [PS]-Stand Down") was highly acceptable to patients, and patients reported significant improvements in drinking outcomes. These data provide a strong foundation for a larger pragmatic trial to test the effectiveness of the Stand Down app and PS-Stand Down to reduce hazardous drinking among Veterans seen in primary care, relative to the current standard of care that these patients receive.

In the current study, the investigators will evaluate whether the Stand Down app reduces drinking among Veteran primary care patients who engage in hazardous drinking, and for whom PS-Stand Down is more effective than the app alone. Aim 1: Test whether Stand Down (vs. Usual Care; UC) and PS-Stand Down (vs. UC and vs. app only) predicts better drinking outcomes, and test mediators of these effects. Aim 2: Test for differences in satisfaction with care across conditions, and conduct qualitative interviews with patients and PACT staff to understand potential barriers/facilitators to implementing PS-Stand Down in primary care. Aim 3: Explore baseline moderators to elucidate for whom PS-Stand Down (vs. app only) is most beneficial.

In a 3-group RCT at the Palo Alto and Syracuse VAs, 274 Veteran primary patients who screen positive for hazardous drinking, received a brief intervention following a positive screen, and are not currently in alcohol use treatment will complete a baseline interview, be randomized to either (i) UC, (ii) UC plus Stand Down, or (iii) UC plus PS-Stand Down (four phone sessions with a Peer over 8 weeks to enhance app engagement), and be re-interviewed at 8, 20, and 32 weeks. For Aim 2, the CFIR framework will guide key informant interviews with 12 patients and 12 PACT providers from each site.

ELIGIBILITY:
Inclusion Criteria:

Veterans will be eligible if they:

* had a positive AUDIT-C screen (score of > 5) during a primary care visit in the past month at a clinic at either the VA Palo Alto Health Care System or the Syracuse VA Medical Center
* have documentation in their medical records of receipt of a BI following a positive screen
* did not receive any outpatient, inpatient, or residential care for alcohol use in the month after their positive AUDIT-C
* own a smartphone

Exclusion Criteria:

* Veterans who have active diagnoses of a psychotic disorder or a cognitive disorder (e.g., dementia) will be excluded
* Veterans who do not agree to be randomized will be excluded as well

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Total standard drinks | 32 weeks post-baseline
  At each assessment, the Timeline Follow Back (TLFB), a retrospective, calendar-based measure, will provide information on quantity/frequency of alcohol use in the past 30 days. Information gathered from this reliable and well-validated measure will be used to calculate total standard drinks

SECONDARY OUTCOMES:
Drinks Per Drinking Day (DPDD) | 32 weeks post-baseline
  At each assessment, the Timeline Follow Back (TLFB), a retrospective, calendar-based measure, will provide information on quantity/frequency of alcohol use in the past 30 days. Information gathered from this reliable and well-validated measure will be used to calculate DPDD.
Heavy Drinking Days (HDD) | 32 weeks post-baseline
  At each assessment, the Timeline Follow Back (TLFB), a retrospective, calendar-based measure, will provide information on quantity/frequency of alcohol use in the past 30 days. Information gathered from this reliable and well-validated measure will be used to calculate HDD (i.e., five or more standard drinks for men and four or more standard drinks for women).
World Health Organization (WHO) drinking risk levels | 32 weeks post-baseline
  At each assessment, the Timeline Follow Back (TLFB), a retrospective, calendar-based measure, will provide information on quantity/frequency of alcohol use in the past 30 days. Information gathered from this reliable and well-validated measure will be used to calculate reductions (one- or two-levels) in WHO drinking risk levels.
Drinks Per Week | 32 weeks post-baseline
  At each assessment, the Timeline Follow Back (TLFB), a retrospective, calendar-based measure, will provide information on quantity/frequency of alcohol use in the past 30 days. Information gathered from this reliable and well-validated measure will be used to calculate drinks per week.
Negative Consequences from Drinking | 32 weeks post-baseline
  The 15-item Short Index of Problems (SIP) will be used to assess negative consequences from drinking. Items are rated on a 4-pt scale (0=Never, 3 = Daily or Almost Daily), which yields a total score.
Percent Days Abstinent (PDA) | 32 weeks post-baseline
  At each assessment, the Timeline Follow Back (TLFB), a retrospective, calendar-based measure, will provide information on quantity/frequency of alcohol use in the past 30 days. Information gathered from this reliable and well-validated measure will be used to calculate PDA.
Self-Efficacy to Reduce Drinking | 32 weeks post-baseline
  Self-efficacy to reduce drinking will be measured at each time point with the 14-item Situational Confidence Questionnaire (SCQ), which asks patients to rate their level of confidence in resisting alcohol use in a range of tempting situations. Responses are rated on a 6-point scale (0%=Not at all confident, 100%=Very confident) are averaged across items to produce a total score, with higher scores indicating more self-efficacy.
Readiness to Change Drinking | 32 weeks post-baseline
  At each time point, the Readiness Ruler will assess patients' readiness to change drinking (quit or cut down). Responses are measured on a 1 (not ready to change) to 10 (trying to change) scale. Higher readiness to change scores predict better alcohol use outcomes in longitudinal studies.
  studies

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Blonigen, PhD MA, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Blonigen DM, Hawkins EJ, Kuhn E, Timko C, Dulin PL, Boothroyd D, Possemato K. Stand Down-Think Before You Drink: protocol for an effectiveness-implementation trial of a mobile application for unhealthy alcohol use with and without peer support. BMJ Open. 2023 Apr 13;13(4):e072892. doi: 10.1136/bmjopen-2023-072892. PMID 37055201

DOCUMENTS (1):
  • Informed Consent Form (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT05473598/ICF_000.pdf